CLINICAL TRIAL: NCT01358552
Title: Néevo®/NéevoDHA® P.L.U.S. Program (Progress Through Learning, Understand & Support)
Status: Terminated | Type: Observational
Why Stopped: Insufficient number of participants
Sponsor: Pamlab, Inc. (Industry)
Collaborators: InfoMedics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: N-003
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Pregnancy
Keywords: Neevo; Neevo DHA; L-methylfolate; anemia during pregnancy; folic acid; vitamin B12; prenatal vitamins; hemoglobin; iron deficiency; Pregnancy
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Néevo®/NéevoDHA®: Subjects who have been prescribed Néevo/NéevoDHA® daily.
  Interventions: Other: Néevo®/ NéevoDHA®

INTERVENTIONS:
Other: Néevo®/ NéevoDHA® — Néevo®/NéevoDHA® is an orally administered medical food indicated for the dietary management of impaired metabolic processes in women under a doctor's care who face high to intermediate risk pregnancies and are unable to fully metabolize or absorb folic acid. Néevo®/ NéevoDHA® contains L-methylfolate, the biologically active and immediately bioavailable form of folate.

SUMMARY:
This is an observational study in which patients who have been prescribed Néevo®/NéevoDHA® are invited to participate in surveys about their pregnancy and experiences with Néevo®/NéevoDHA®. The purpose of this study is to increase the understanding of the role of L-methylfolate among patients who are candidates for Néevo®/NéevoDHA®, provide patients with personalized education and support during their pregnancies, and contribute to the overall understanding of the needs and concerns of women facing intermediate- to high-risk pregnancies.

DETAILED DESCRIPTION:
Surveys used to conduct this study will be administered via telephone or online by InfoMedics, Inc., a company with a system for developing such patient-physician feedback programs. Participating physicians will ask their patients to participate in the program after Néevo®/NéevoDHA® has been prescribed and provide them with a patient brochure containing an introduction to the program and instructions on how to enroll. Patients interested in participating self-enroll, take a brief survey before starting their Néevo®/NéevoDHA® prescription, and then a follow-up survey 4 weeks after they have started taking Néevo®/NéevoDHA®. As patients complete surveys within the study, their physician will receive individualized feedback reports outlining their patient's treatment experience and progress. Patients will also receive a copy of their own reports, to help encourage them to continue taking Néevo®/NéevoDHA® as directed. Patients will also receive educational materials about diet and nutrition during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* New Néevo®/NéevoDHA® Start.
* Only for women who are pregnant and taking brand name Néevo®/ NéevoDHA® under a physicians care.

Exclusion Criteria:

* Patients who are not pregnant.
* If participant indicates that she did not get a prescription for Néevo®/ NéevoDHA®, she will not be able to complete the survey(s).
* For the follow-up survey, if the participant indicates that she has not been taking Néevo®/NéevoDHA®, she will not be able to complete the survey( (s).

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who have been prescribed Néevo®/ NéevoDHA®
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of Néevo®/NéevoDHA® as measured by side effects and compliance | Week 4
  To collect data from patient surveys on the patient utilization and effectiveness of Néevo®/NéevoDHA® in a "real world" setting.

SECONDARY OUTCOMES:
To determine overall patient satisfaction with Néevo®/NéevoDHA® using a 9-point satisfaction scale | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Noe Lira, M.D., Principal Investigator — Noe Lira, M.D.
Locations (1):
- Noe Lira, M.D., Corpus Christi, Texas, United States